CLINICAL TRIAL: NCT05822752
Title: A Phase 2, Randomized Study to Evaluate the Optimized Dose, Safety, and Efficacy of Livmoniplimab in Combination With Budigalimab for Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC) Patients Who Have Progressed After an Immune Checkpoint Inhibitor Containing Regimen in First-Line HCC
Brief Title: Study to Evaluate Adverse Events, and Change in Disease Activity, When Intravenously (IV) Infused With Livmoniplimab in Combination With IV Infused Budigalimab in Adult Participants With Hepatocellular Carcinoma (HCC)
Acronym: LIVIGNO-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M24-147; 2022-502948-13-00 (Other: EU CT)
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; Sorafenib; Livmoniplimab; Budigalimab; ABBV-181; ABBV-151; Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms | interventions — budigalimab; lenvatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: Lenvatinib or Sorafenib (Active Comparator): Participants will receive Lenvatinib or or Sorafenib, as part of an approximately 2 year treatment period.
  Interventions: Drug: Lenvatinib; Drug: Sorafenib
- Arm 2: Livmoniplimab Dose A + Budigalimab (Experimental): Participants will receive Livmoniplimab Dose A in combination with budigalimab, as part of an approximately 2 year treatment period.
  Interventions: Drug: Budigalimab; Drug: Livmoniplimab
- Arm 3: Livmoniplimab Dose B + Budigalimab (Experimental): Participants will receive Livmoniplimab Dose B in combination with budigalimab, as part of an approximately 2 year treatment period.
  Interventions: Drug: Budigalimab; Drug: Livmoniplimab

INTERVENTIONS:
Drug: Budigalimab — Intravenous (IV) Infusion
  Other Names: ABBV-181
  Arms: Arm 2: Livmoniplimab Dose A + Budigalimab; Arm 3: Livmoniplimab Dose B + Budigalimab
Drug: Livmoniplimab — Intravenous (IV) Infusion
  Other Names: ABBV-151
  Arms: Arm 2: Livmoniplimab Dose A + Budigalimab; Arm 3: Livmoniplimab Dose B + Budigalimab
Drug: Lenvatinib — Oral: Capsule
  Arms: Arm 1: Lenvatinib or Sorafenib
Drug: Sorafenib — Oral: Tablet
  Arms: Arm 1: Lenvatinib or Sorafenib

SUMMARY:
Hepatocellular carcinoma (HCC) is a common cancer worldwide and a leading cause of cancer-related death. The majority of participants first presenting with HCC have advanced unresectable or metastatic disease. The purpose of this study is to evaluate the optimized dose, adverse events, and efficacy of livmoniplimab in combination with budigalimab.

Livmoniplimab is an investigational drug being developed for the treatment of HCC. There are 3 treatment arms in this study and participants will be randomized in a 1:1:1 ratio. Participants will either receive livmoniplimab (at different doses) in combination with budigalimab (another investigational drug), lenvatinib, or sorafenib. Approximately 120 adult participants will be enrolled in the study across 60 sites worldwide.

In arm 1 (control), participants will receive the investigator's choice: lenvatinib as an oral capsule or sorafenib as an oral tablet, once daily. In arm 2, participants will receive intravenously (IV) infused livmoniplimab (dose A) in combination with IV infused budigalimab, every 3 weeks. In arm 3, participants will receive intravenously (IV) infused livmoniplimab (dose B) in combination with IV infused budigalimab, every 3 weeks. The estimated duration of the study is up to 2 years

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, questionnaires, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh A classification.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Received an immune checkpoint inhibitor in first-line (1L) hepatocellular carcinoma (HCC) treatment regimen.
* Adequate hematologic and end-organ function.
* Tissue biopsy at screening.
* Disease that is not amenable to surgical and/or locoregional therapies, or progressive disease after surgical and /or locoregional therapies.

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.
* Prior treatment with an approved tyrosine kinase inhibitor (for example sorafenib or Lenvatinib) in 1L HCC treatment regimen.
* History of malignancy other than hepatocellular carcinoma (HCC) within 5 years prior to screening.
* Hepatic encephalopathy or requirement for medications to prevent or control encephalopathy.
* Moderate or severe ascites requiring recurrent non-pharmacologic intervention to maintain symptomatic control.
* Coinfection with active HBV infection and active HCV infection.
* Prior history of grade 3 or higher immune-mediated adverse event or discontinuation due to immune-mediated adverse events.
* Prior history of recurrent grade 2 or higher interstitial lung disease/pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response (BOR) per Investigator | Through Study Completion, Up to Approximately 27 Months
  BOR is defined as a subject achieving confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as determined by investigators at any time prior to subsequent anticancer therapy.

SECONDARY OUTCOMES:
Duration of response (DOR) per Investigator | Through Study Completion, Up to Approximately 27 Months
  DOR is defined as the time from first confirmed CR or PR until the first documentation of progressive disease according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.
Number of Participants with Progression-free Survival (PFS) | Through Study Completion, Up to Approximately 27 Months
  PFS is defined as the time from randomization until the first documentation of progressive disease according to RECIST 1.1 as determined by investigators or death from any cause, whichever occurs first.
Overall Survival (OS) | Through Study Completion, Up to Approximately 27 Months
  OS is defined as the time from randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (59):
- United States (20):
  - Arizona Oncology Associates, PC - NAHOA Prescott Valley /ID# 254313, Prescott Valley, Arizona
  - Highlands Oncology Group, PA /ID# 253158, Springdale, Arkansas
  - University of California, Los Angeles /ID# 253292, Los Angeles, California
  - UC Irvine /ID# 252707, Orange, California
  - California Pacific Medical Center - San Francisco - Webster Street /ID# 253291, San Francisco, California
  - Rocky Mountain Cancer Centers - Denver Midtwon /ID# 254163, Denver, Colorado
  - AdventHealth Orlando /ID# 252865, Orlando, Florida
  - The University of Chicago Medical Center /ID# 252870, Chicago, Illinois
  - Hematology/Oncology Clinic /ID# 253851, Baton Rouge, Louisiana
  - Dana-Farber Cancer Institute /ID# 252696, Boston, Massachusetts
  - Henry Ford Hospital /ID# 253342, Detroit, Michigan
  - Washington University-School of Medicine /ID# 252698, St Louis, Missouri
  - NYU Langone - Laura and Isaac Perlmutter Cancer Center /ID# 252708, New York, New York
  - Memorial Sloan Kettering Cancer Center-Koch Center /ID# 252705, New York, New York
  - Messino Cancer Center - Asheville /ID# 253888, Asheville, North Carolina
  - University of North Carolina /ID# 252739, Chapel Hill, North Carolina
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 252699, Providence, Rhode Island
  - Duplicate_Texas Oncology - Medical City Dallas /ID# 254164, Dallas, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 252770, Dallas, Texas
  - Texas Oncology - Northeast Texas /ID# 254184, Tyler, Texas
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux /ID# 252749, Pessac, Gironde
  - CHU Montpellier - Hopital Saint Eloi /ID# 252760, Montpellier, Herault
  - CHU Grenoble - Hopital Michallon /ID# 252755, La Tronche, Isere
  - CHRU Lille - Hopital Claude Huriez /ID# 252748, Lille, Nord
  - AP-HP - Hopital Paul-Brousse /ID# 253646, Villejuif
  - Hopital Beaujon /ID# 252758, Clichy, Île-de-France Region
- Italy (6):
  - Azienda Ospedaliero Universitaria Careggi /ID# 254444, Florence, Firenze
  - IRCCS Ospedale San Raffaele /ID# 252910, Milan, Milano
  - P.O. Ospedale del Mare /ID# 253140, Naples, Napoli
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 253247, Bologna
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 253142, Palermo
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 253141, Roma
- Japan (5):
  - Chiba University Hospital /ID# 255190, Chiba, Chiba
  - National Cancer Center Hospital East /ID# 253419, Kashiwa-shi, Chiba
  - Kanazawa University Hospital /ID# 254861, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center /ID# 255790, Yokohama, Kanagawa
  - Kindai University Hospital /ID# 255106, Osakasayama-shi, Osaka
- South Korea (5):
  - CHA Bundang Medical Center /ID# 253054, Seongnam, Gyeonggido
  - Seoul National University Bundang Hospital /ID# 253412, Seongnam-si, Gyeonggido
  - Chonnam National University Hwasun Hospital /ID# 253133, Hwasun-gun, Jeonranamdo
  - Asan Medical Center /ID# 253044, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 253411, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Hospital Universitario Marques de Valdecilla /ID# 253059, Santander, Cantabria
  - Hospital Universitario Reina Sofia /ID# 253083, Córdoba, Cordoba
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 253078, Majadahonda, Madrid
  - Clinica Universidad de Navarra - Pamplona /ID# 253073, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron /ID# 253063, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 254840, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 253074, Seville
  - Hospital Universitario Miguel Servet /ID# 253071, Zaragoza
- Taiwan (9):
  - E-DA Cancer Hospital /ID# 260881, Kaohsiung City, Kaohsiung
  - Kaohsiung Chang Gung Memorial Hospital /ID# 253675, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 253449, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 253451, Kaohsiung City
  - China Medical University Hospital /ID# 253453, Taichung
  - Taichung Veterans General Hospital /ID# 253452, Taichung
  - National Cheng Kung University Hospital /ID# 253676, Tainan
  - Taipei Veterans General Hosp /ID# 253450, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 253674, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info. — https://www.abbvieclinicaltrials.com/study/?id=M24-147